CLINICAL TRIAL: NCT00000227
Title: Alternate-Day Buprenorphine Administration. Phase VIII
Brief Title: Alternate-Day Buprenorphine Administration. Phase VIII - 9
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Model: Crossover | Purpose: Treatment
Other Study IDs: NIDA-06969-9; R01DA006969 (NIH); R01-06969-9
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 1996-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate open buprenorphine dosing with dose choice.

ELIGIBILITY:
Please contact site for information.

Ages: 25 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-08

PRIMARY OUTCOMES:
Drug use
Opioid withdrawal
Opioid agonist effects
Dose choice

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States